CLINICAL TRIAL: NCT04676919
Title: Phonophoresis Therapy in Subacromial Impingement Syndrome: Comparing of Pulsed Mode Ultrasound Phonophoresis and Continuous Mode Ultrasound Phonophoresis.
Brief Title: The Effect of Phonophoresis in Subacromial Impingement Syndrome.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Volkan Deniz, PT, MSc, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 72/1185
Record Dates: First submitted 2020-12-18; First posted 2020-12-21 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Subacromial Impingement Syndrome
Keywords: subacromial pain; ultrasound therapy; phonophoresis
MeSH Terms: conditions — Shoulder Impingement Syndrome | interventions — Phonophoresis

STUDY DESIGN:
Who Masked: Participant
Masking Description: sham
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- pulsed mode phonophoresis group (Experimental): Phonophoresis therapy with pulsed mode ultrasound.
  Interventions: Device: phonophoresis therapy with pulsed mode ultrasound
- continuous mode phonophoresis group (Experimental): Phonophoresis therapy with continuous mode ultrasound.
  Interventions: Device: phonophoresis therapy with continuous mode ultrasound
- sham group (Sham Comparator): Sham ultrasound
  Interventions: Device: sham ultrasound

INTERVENTIONS:
Device: phonophoresis therapy with pulsed mode ultrasound — phonophoresis therapy with pulsed mode ultrasound, five days a week for three weeks
  Arms: pulsed mode phonophoresis group
Device: phonophoresis therapy with continuous mode ultrasound — phonophoresis therapy with pulsed mode ultrasound, five days a week for three weeks
  Arms: continuous mode phonophoresis group
Device: sham ultrasound — sham ultrasound therapy, five days a week for three weeks
  Arms: sham group

SUMMARY:
Subacromial impingement syndrome (SIS) is a dysfunction caused by an impingement of the rotator cuff tendon between the head of the humerus and the acromion as a result of changes in the subacromial space. The patients' symptoms, such as pain, limited joint mobility and reduced strength, may lead to a diagnosis of SIS. The conservative treatment of individuals with SIS is includes analgesics and non-steroidal anti-inflammatory drugs (NSAIDs), steroid injections and physiotherapy. Ultrasound therapy is one of the common physiotherapy applications for SIS, but its effectiveness is controversial. Phonophoresis is a combination of ultrasound therapy and medical therapy. In phonophoresis, a medicine in gel form is used as a transmitter with ultrasound instead of the aquatic conductor gel. It was hypothesized that ultrasound waves favoring the penetration of an anti-inflammatory drug would lead to an improved response to the treatment of SIS. However, the effectiveness of ultrasound modes (pulsed or continuous) can be used in phonophoresis is debatable. The purpose of this study is to determine the effect of ultrasound therapy, pulsed mode ultrasound and continuous mode ultrasound phonophoresis in patients with SIS.

ELIGIBILITY:
Inclusion Criteria:

* to be diagnosed as shoulder impingement syndrome,
* shoulder pain for at least one month,
* VAS score over 40mm.

Exclusion Criteria:

* grade III supraspinatus tendon injury,
* major shoulder trauma,
* diabetes mellitus,
* hipotiroidizm,
* adhesive capsulitis,
* cardiac pacemaker
* physical therapy or local injection to the shoulder at last six month
* serious cervical pathologies.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2021-01-15 (Actual); Study Completion 2021-01-30 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale | Baseline, Change from baseline pain scores at three weeks, Change from baseline pain scores at three months
  The visual analog scale (VAS) is a pain rating scale first used by Hayes and Patterson in 1921. Scores are based on self-reported measures of symptoms that are recorded with a single handwritten mark placed at one point along the length of a 10-cm line that represents a continuum between the two ends of the scale-"no pain" on the left end (0 cm) of the scale and the "worst pain" on the right end of the scale (10 cm).
The Shortened version of Disability of the Arm, Shoulder, and Hand | Baseline, Change from baseline shoulder pain and function scores at three weeks, Change from baseline shoulder pain and function at three months
  Disability of the Arm, Shoulder, and Hand (DASH) was designed to describe disability experienced by patients with any musculoskeletal condition of the upper extremity and to monitor change in symptoms and upper limb function over time. The DASH questionnaire has been validated in patients with upper extremity musculoskeletal disorders such as rheumatoid arthritis and shoulder impingement syndrome. The Quick-DASH is a shortened version of the DASH

SECONDARY OUTCOMES:
Nottingham Health Profile | Baseline, Change from baseline quality of life scores at three weeks, Change from baseline quality of life scores at three months
  Nottingham Health Profile (NHP) evaluates emotional, social, and physical health problems perceived by the patient. It consists of six parts: pain (8 items), emotional reactions (9 items), sleep (5 items), social isolation (5 items), physical mobility (8 items), and energy level (3 items). Higher scores correspond to poorer perceived health status.

CONTACTS AND LOCATIONS:
Overall Officials: Bayram Kelle, Assoc. Prof., Principal Investigator — Cukurova University
Locations (1):
- Volkan deniz, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No